CLINICAL TRIAL: NCT06747455
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase III Clinical Trial Evaluating the Efficacy and Safety of Therapeutic BCG for the Prevention of Postoperative Recurrence of Non-muscle-invasive Bladder Cancer in People Aged 18 Years and Older
Brief Title: BCG for Therapeutic Use Phase Ⅲ Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LKM-2024-BCG01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: BCG
Keywords: Bacillus Calmette-Guérin for treatment; Bladder cancer.
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Therapeutic Uses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Common name: BCG for Therapeutic Use Specification: 60mg/bottle. Each bottle contains 60mg of BCG, and the number of viable bacteria per 1mg BCG should not be less than 1.0×10^6CFU.
  Expiration date: 24 months. Production unit: Anhui Zhifeilong Kema Biopharmaceutical Co., Ltd.
  Interventions: Drug: BCG for Therapeutic Use
- Control group (Active Comparator): Common name: BCG for Therapeutic Use ( BI SAI JI ) Specification: 60mg (6.0×10^7CFU)/bottle. Each bottle contains 60mg of BCG, and the number of viable bacteria per 1mg BCG should not be less than 1.0×10^6CFU.
  Expiration date: 18 months. Production unit: Chengdu Institute of Biological Products Co., Ltd.
  Interventions: Drug: BCG for Therapeutic Use ( BI SAI JI )

INTERVENTIONS:
Drug: BCG for Therapeutic Use — After the subjects after transurethral bladder tumor resection were screened and randomly enrolled, the subjects were given intravesical infusion (experimental drug) within 2~12 weeks after surgery, and perfused once a week for 6 consecutive times during the induction period; During the intensive phase, perfusion is given once every two weeks, 3 times in a row; During the maintenance period, perfusion was given once every 4 weeks, for a total of 19 perfusions, and the perfusion time continued until 1 year after surgery.
  Arms: Experimental group
Drug: BCG for Therapeutic Use ( BI SAI JI ) — After the subjects after transurethral bladder tumor resection were screened and randomly enrolled, the subjects were administered intravesical infusion (control drug) within 2~12 weeks after surgery, and perfused once a week for 6 consecutive times during the induction period; During the intensive phase, perfusion is given once every two weeks, 3 times in a row; During the maintenance period, perfusion was given once every 4 weeks, for a total of 19 perfusions, and the perfusion time continued until 1 year after surgery.
  Arms: Control group

SUMMARY:
Research topic: A randomized, double-blind, active-controlled, multicenter phase III clinical trial evaluating the efficacy and safety of therapeutic BCG for the prevention of postoperative recurrence of non-muscle-invasive bladder cancer in people aged 18 years and older.

The name of the drug: Bacillus Calmette-Guérin for treatment(BCG). Clinical indications: It is used for the treatment of bladder carcinoma in situ and the prevention of recurrence, and for the prevention of recurrence of bladder papilloma after transurethral resection in Ta or T1 stage. This product is not used for papillomas beyond the T1 stage.

Study population: Patients aged 18 years and above with intermediate- and high-risk non-muscle-invasive bladder cancer (NMIBC) who have undergone transurethral bladder tumor resection.

Objectives: Primary Objectives: To assess the effectiveness of BCG for therapeutic use in the adjuvant treatment of intermediate- and high-risk NMIBC after transurethral resection of bladder tumors. Secondary Purpose: To assess the safety of the therapeutic BCG vaccine in the adjuvant treatment of intermediate- and high-risk NMIBC after transurethral resection of bladder tumors. Other purposes: To assess the pharmacodynamic (PD) profile of BCG for therapeutic use in the adjuvant treatment of intermediate- and high-risk NMIBC after transurethral resection of bladder tumors.

Study design: This study adopts a randomized, double-blind, active-controlled, multi-center trial design, including three phases: screening period, treatment period and follow-up period. In this study, 438 subjects will be randomly assigned to the experimental group and the control group in a 1:1 ratio, with 219 patients in both the experimental group and the control group, and stratified according to the baseline risk level (high-risk/intermediate-risk) and whether or not to perform urine PD sample collection (yes/no).

DETAILED DESCRIPTION:
Research topic: A randomized, double-blind, active-controlled, multicenter phase III clinical trial evaluating the efficacy and safety of therapeutic BCG for the prevention of postoperative recurrence of non-muscle-invasive bladder cancer in people aged 18 years and older.

Study endpoints: Endpoint efficacy: Main efficacy measures: 1-year recurrence-free survival rate (1-year RFS%): To assess the proportion of participants who are relapse-free or die from randomization up to 1 year, whichever occurs first. Secondary efficacy endpoint: 2-year recurrence-free survival rate (2-year RFS%): Assessing the proportion of subjects who have not experienced recurrence or death (whichever occurs first) from randomization until 2 years. 1-year progression-free survival rate (1-year PFS%): Assessing the proportion of subjects experiencing tumor progression or death from randomization until 1 year. The 2-year progression-free survival rate (2-year PFS%) assesses the proportion of subjects experiencing tumor progression or death from the time of randomization until 2 years. Security endpoint: Incidence of all AEs and SAEs; Any clinically significant abnormalities in vital signs or physical examinations during the trial period; Any clinically significant abnormalities found during the trial period laboratory examinations or electrocardiogram examinations. Other destinations: Changes in the levels of interleukin 2 (IL-2), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-12 (IL-12), interferon γ (IFN-γ), and tumor necrosis factor (TNF) in urine excreted at 4 h±1 h, 8 h±, 2 h, and 24 h±3 h after the 1st (V1), 6th (V6), 9th (V9), and 10th (V10) administration.

Overall design: This study adopts a randomized, double-blind, positive-controlled, multicenter trial design, including three phases: screening, treatment, and follow-up. A total of 438 subjects will be enrolled in this study, with a 1:1 random allocation to the experimental group and the control group, both consisting of 219 subjects. Stratification will be based on baseline risk level (high risk/medium risk) and whether urine PD samples are collected (yes/no). Selection period: During the first 28 days prior to administration, the subjects will undergo eligibility confirmation for enrollment. Subjects who meet the eligibility criteria will enter the treatment phase and receive the investigational drug infusion.

Treatment period (Year 1): The treatment period includes the induction phase, consolidation phase, and maintenance phase.

After undergoing transurethral bladder tumor resection, eligible subjects are screened and randomly assigned to the study. Within 2 to 12 weeks after surgery, subjects receive bladder instillation therapy: once a week during the induction phase for a total of 6 times, once every two weeks during the consolidation phase for a total of 3 times, and once every 4 weeks during the maintenance phase for a total of 19 times, continuing until 1 year after surgery.

During the first year of the study, subjects undergo imaging examinations every 12 months, urine cytology examinations every 3 months, and cystoscopy. If a subject shows positive results in either cystoscopy or urine cytology, the researcher may decide to perform additional imaging examinations.

Early Termination of Treatment Visit: For subjects who discontinue treatment early without completing the first year of infusion therapy in the treatment period and without experiencing tumor recurrence or progression, an Early Termination of Treatment Visit will be conducted within 30 days after the last dose. If subsequent other local or systemic anti-tumor therapies are received, this should be accurately recorded.

Follow-up period (Year 2): After completing the first year of infusion therapy in the treatment period, or for subjects who discontinued treatment early without tumor recurrence or progression, or subjects who continue receiving treatment into the second year, follow-up will be conducted during the second year of the study. All subjects meeting the above conditions will undergo imaging examinations every 12 months, and urine cytology examinations and cystoscopy every 3 months, until the subject experiences tumor recurrence or progression, withdraws informed consent, is lost to follow-up, the sponsor terminates the study, or death occurs (whichever occurs first). If a subject has a positive result in either cystoscopy or urine cytology, the investigator may decide to perform additional imaging examinations.

This trial plans to conduct the first analysis of the efficacy and safety of the investigational product after all subjects have experienced recurrence or death, or have completed one year of follow-up observation. The first analysis will involve unblinding and statistical analysis performed by a firewalled unblinded team, while the main study team will remain blinded at the individual subject level to continue follow-up of trial subjects. The final unblinding and statistical analysis will be conducted upon completion of the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age≥ 18 years old, male or female;
* 2. According to the Guidelines for the Diagnosis and Treatment of Bladder Cancer (2022 Edition), the initial histological diagnosis of intermediate- and high-risk non-muscle-invasive urothelial carcinoma of the bladder (T1, Ta or Tis) and the need for BCG bladder infusion adjuvant therapy is evaluated;
* 3. Patients undergoing transurethral bladder tumor resection need to meet the requirements of all tumors to have no visible tumors after surgery. This study can also enroll patients who need a second electroresection, subjects who meet the secondary electroresection criteria are recommended to undergo secondary electroresection and should be included in the study after comprehensive evaluation based on the two pathological results (BCG perfusion for treatment should be carried out within 2~12 weeks after surgery, cystoscopy should be added more than 4 weeks after surgery to ensure that there is no visible tumor after surgery, and the subjects who underwent secondary resection should be calculated based on the postoperative time of the second electroresection); Note: The criteria for the second resection: (1) the first TURBt is insufficient; (2) the first electrosection of non-myometrial tissue specimens; (3) T1 tumors; (4) High-grade (G3) tumors, except for carcinoma in situ. The second resection is recommended to be performed within 2-6 weeks after the first resection, and no other perfusion therapy is allowed except for the bladder infusion chemotherapy drugs immediately after the first and second resection;
* 4. Eastern Cooperative Oncology Group (ECOG) score (see Appendix 1 for details): 0~2 points;
* 5. At screening, clinical laboratory tests meet the following characteristics:

  1. Blood routine: no use of hematopoietic growth factors or blood transfusion support within 14 days before randomization, including: absolute neutrophil count (ANC) ≥1500/mm^3 or ≥1.5×10^9/L; Platelets≥ 100000/mm^3 or 100×10^9/L; Hemoglobin ≥ 9 g/dL.
  2. Liver function: total bilirubin ≤ 1.5× upper limit of normal range (ULN), subjects with Gilbert's syndrome require total bilirubin <3×ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN.
  3. Renal function: defined as creatinine clearance estimated according to the Cockcroft Gault formula (Appendix 2) ≥ 30mL/min;
  4. Coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5×ULN, and the international normalized ratio (INR) ≤ 1.5×ULN.
* 6. Voluntarily participate in this trial, with full informed consent and signed written informed consent.

Exclusion Criteria:

* 1. Those who have immunodeficiency or damage (such as AIDS patients), are using immunosuppressive drugs, steroid hormones, etc., which may cause systemic BCG disease reaction (other hormones such as patients who are given corresponding hormone therapy after thyroid/adrenal resection can be enrolled);
* 2. Those who are allergic to BCG and its excipients;
* 3. Active tuberculosis, those who are receiving or have received anti-tuberculosis treatment within 6 months before screening;
* 4. Patients with severe cardiovascular and cerebrovascular, liver, lung, and kidney diseases at the time of screening;
* 5. Patients with urothelial carcinoma or other urogenital tumors or other organ tumors in any part outside the bladder during screening, and no obvious tumor recurrence or progression in the past 3 years, and stable condition can be considered for inclusion, such as basal cell or squamous cell skin cancer that has been adequately treated; carcinoma in situ of the breast or cervix; Low-grade prostate cancer that is monitored without any planned therapeutic intervention (e.g., surgery, radiotherapy, or castration); and other concurrent malignancies that in the opinion of the investigator have a very low likelihood of progression;
* 6. Patients with histologically confirmed muscle-invasive, locally advanced, unresectable or metastatic urothelial carcinoma or a history of this disease (i.e., ≥ T2);
* 7. Those who have received any BCG treatment for NMIBC in the past;
* 8. Those who know or suspect that abnormal conditions such as bladder perforation occur during surgery;
* 9. Those who suspect that the surgical wound has not healed or the urinary tract mucosa is damaged;
* 10. Those who have been assessed by the investigator to be accompanied by cystitis (such as urinary frequency, urgency, dysuria, etc.), or have received other bladder infusion drugs and have severe bladder irritation, which is expected to affect the evaluation of this study;
* 11. In addition to immediate postoperative intravesical chemotherapy, patients who have received other systemic anti-tumor treatments such as chemotherapy, radiotherapy, and immunotherapy for the disease under study;
* 12. Pregnant or lactating women;
* 13. Those who cannot guarantee effective contraception during the trial period to 6 months after the last dose;
* 14. Received treatment with other clinical trial drugs (except placebo) or clinical trial devices within 3 months before the first dose;
* 15. Those who have a history of alcoholism, drug abuse or drug abuse within 6 months before screening;
* 16. Presence of any of the following: positive human immunodeficiency virus (HIV) antibody, positive syphilis-specific antibody, active hepatitis B (hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (DNA) copy number ≥200 IU/mL or 1000 copies/mL), hepatitis C virus (HCV) antibody positive and HCV virus copy number higher than the upper limit of normal in the research center≥ 10^3/mL;
* 17. Any condition that, in the opinion of the investigator, may increase the risk of the subject or interfere with the performance of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year RFS% | Up to 1 year after randomization
  To assess the proportion of participants who were free of recurrence or death (whichever occurs first) from randomisation up to 1 year.
Safety endpoints | 30 days after the last dose
  Incidence of all AEs
Safety endpoints | 30 days after the last dose
  Incidence of all SAEs
Safety endpoints | 30 days after the last dose
  Any clinically significant abnormalities of vital signs during the trial
Safety endpoints | 30 days after the last dose
  Any clinically significant abnormalities found in the physical examination during the trial
Safety endpoints | 30 days after the last dose
  Any clinically significant abnormalities in laboratory tests during the trial
Safety endpoints | 30 days after the last dose
  Any clinically significant abnormalities in the electrocardiogram (ECG) examination during the trial

SECONDARY OUTCOMES:
2-years RFS% | Up to 2 years after randomization
  To assess the proportion of participants who were free of recurrence or death (whichever occurs first) from randomization up to 2 years.
1-year PFS% | Up to 1 year after randomization
  To assess the proportion of participants with tumor progression or death from randomization up to 1 year.
2-years PFS% | Up to 2 years after randomization
  To assess the proportion of participants with tumour progression or death from randomisation up to 2 years.

OTHER OUTCOMES:
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of IL-2 in urine
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of IL-6 in urine
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of IL-8 in urine
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of IL-12 in urine
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of IFN-γ in urine
To evaluate the PD characteristics of the therapeutic BCG vaccine for adjuvant therapy after transurethral resection of intermediate- and high-risk NMIBC | The 1st , 6th , 9th and 10th (V10) doses were last excreted before administration, 4 h±1 h, 8 h± 2 h, and 24 h±3 h after administration
  Changes in levels of TNF in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China